CLINICAL TRIAL: NCT07312331
Title: SOC-based Behavioral Intervention to Promote Walking and Well-being Among Older Adults in Jiazhou, China
Brief Title: SOC-based Behavioral Intervention to Promote Walking
Acronym: SOCWalk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ling Yang (Other)
Responsible Party: Sponsor-Investigator, Ling Yang, Ph.D., Chinese University of Hong Kong
Organization: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: SOCWALK2025
Record Dates: First submitted 2025-11-25; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Older Adults; Older Adults (65 Years and Older)
Keywords: Selection, Optimization, and Compensation (SOC); walking behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SOC (Experimental): SOC-based walking intervention
  Interventions: Behavioral: SOC-based walking intervention
- Active control group (Active Comparator): active health education control.
  Interventions: Other: general health education program

INTERVENTIONS:
Behavioral: SOC-based walking intervention — A structured Selection, Optimization, and Compensation (SOC)-based workshop designed to promote adaptive self-regulation in the domain of physical activity, particularly walking
  Arms: SOC
Other: general health education program — A general health education program that covered age-related topics such as nutrition, sleep, medication adherence, and mental well-being, but excluded any self-regulatory or goal-setting components.
  Arms: Active control group

SUMMARY:
Drawing on the Selection, Optimization, and Compensation (SOC) model of adaptive development, this study tested whether a structured behavioral intervention could enhance walking activity and well-being through improvements in self-regulatory strategy use.

ELIGIBILITY:
Inclusion Criteria:

* Individuals were excluded if they had moderate-to-severe cognitive impairment, medical contraindications for walking, or planned relocation within six months.

Exclusion Criteria:

* Eligible participants were Chinese adults aged 65 years or older, lived in urban areas, could walk independently for at least 10 minutes, and had access to a mobile phone or WeChat (personally or through a family member).

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 350 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Walking behavior | From enrollment to the end of treatment at 8 weeks
  weekly minutes of walking

SECONDARY OUTCOMES:
Selection | From enrollment to the end of treatment at 8 weeks
  Use of "SOC (Selection, Optimization, and Compensation strategies)" questionnaire specific to walking, assessed with brief subscales (3-4 items each; 5-point Likert), at T0, T1, and T2. It assesses the self-regulatory strategies using a 12-item version of the Selection Questionnaire originally developed by Freund and Baltes (2002) and validated for use with Chinese older adults by Chou and Chi (2001). The instrument comprises three subscales-in this case we use the Selection scale-with four items rated on a 5-point Likert scale (1 = strongly disagree, 5 = strongly agree).
Optimization | From enrollment to the end of treatment at 8 weeks
  Use of SOC "Selection, Optimization, and Compensation strategies Questionnaire" specific to walking, assessed with brief subscales (3-4 items each; 5-point Likert), at T0, T1, and T2. For this outcome, we use the subscale Optimization, which self-regulatory strategies assessed using a list of Optimization items, originally developed by Freund and Baltes (2002) and validated for use with Chinese older adults by Chou and Chi (2001). The instrument comprises is rated on a 5-point Likert scale (1 = strongly disagree, 5 = strongly agree).
Compensation | From enrollment to the end of treatment at 8 weeks
  Use of SOC "Selection, Optimization, and Compensation strategies Questionnaire" specific to walking, assessed with brief subscales (3-4 items each; 5-point Likert), at T0, T1, and T2. We use the Compensation subscale of self-regulatory strategies, that was originally developed by Freund and Baltes (2002) and validated for use with Chinese older adults by Chou and Chi (2001). The instrument is rated on a 5-point Likert scale (1 = strongly disagree, 5 = strongly agree).

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Polytechnic University, Jiaozuo, Henan, China

IPD SHARING:
Plan to Share IPD: No
The protection of the privacy of our respondents does not allow us to share IPD.